CLINICAL TRIAL: NCT01689194
Title: A Phase II Study of Genexol-PM and Cisplatin as Induction Chemotherapy in Unresectable, Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Efficacy Study of Genexol-PM and Cisplatin in Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Clinical Research Center for Solid Tumor, Korea (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L-0007; H-1204-103-407 (Other: SNUH IRB)
Record Dates: First submitted 2012-08-30; First posted 2012-09-21 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin

ARMS (1):
- genexolPM + cisplatin (Experimental)
  Interventions: Drug: genexolPM + cisplatin

INTERVENTIONS:
Drug: genexolPM + cisplatin

SUMMARY:
This clinical trial is Phase II trial for evaluating efficacy of induction chemotherapy using Genexol-PM + cisplatin for locally advanced head and neck cancer. The investigators try to evaluate response rate of Genexol-PM + cisplatin chemotherapy, and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced head and neck squamous cell carcinoma
* oral cavity, oropharynx, hypopharynx, larynx
* measurable lesion
* unresectable
* age 18 or more
* ECOG 0 or 1

Exclusion Criteria:

* distant metastasis
* pregnancy
* prior chemotherapy or radiation therapy
* 2ndary malignancy
* other unfit medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
response rate | every 2 cycles, 6wk later after chemotherapy
  RECIST

SECONDARY OUTCOMES:
Locoregional control rate | every 3wk (every cycle)
  NCI CTCAE
Quality of life | every 3wk (every cycle)
  EORTC Q30; performance scale(activities) pain adverse event(appetite, sleep and so on)
safety | every 3wk (every cycle)
  NCI CTCAE v3.0; disease or syndrome, pathologic funtion, sign or symptom, imjury or poisoning, anatomical abnormality, mental or behavioral dysfunction Neutropenia, leucopenia, thrombocytopenia, hepatotoxicity, renal toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Keam B, Lee KW, Lee SH, Kim JS, Kim JH, Wu HG, Eom KY, Kim S, Ahn SH, Chung EJ, Kwon SK, Jeong WJ, Jung YH, Kim JW, Heo DS. A Phase II Study of Genexol-PM and Cisplatin as Induction Chemotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma. Oncologist. 2019 Jun;24(6):751-e231. doi: 10.1634/theoncologist.2019-0070. Epub 2019 Feb 22. PMID 30796155